CLINICAL TRIAL: NCT07191496
Title: Quality of Life in Breast Cancer Survivors Who Were Pregnant During Their Cancer Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-0909; NCI-2025-06866 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2025-09-16; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Survivor; Pregnant Women; Quality of Lifte
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire — The questionnaires include the Ferrans and Powers QLI, EORTC QLQ-C30, FCR-7 Scale, HADS, and MOS Social Support Survey.

SUMMARY:
To assess the quality of life for women who were pregnant during their breast cancer treatment.

DETAILED DESCRIPTION:
Primary Objectives Provide preliminary data to describe the current QOL of breast cancer survivors who received cancer treatment while pregnant.

Secondary Objectives Identify the relationship between QOL and anxiety, depression, fear of cancer recurrence, and social support in breast cancer survivors, who received treatment while pregnant.

ELIGIBILITY:
Eligibility Criteria

* Female, any current age and any age at diagnosis
* Documented diagnosis of breast cancer during pregnancy
* Documentation of receiving chemotherapy during pregnancy
* Alive with no evidence of disease at time of recruitment
* Able to reach and speak English

Exclusion Criteria

* Any woman who delayed and received their chemotherapy after delivery.
* Any woman who was diagnosed with breast cancer before or after their pregnancy.
* Any woman whom there is documentation of inability to provide consent in the medical record

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Females
Study Population: MD Anderson Cancer Center
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-22 (Estimated); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
QOL Questionnaires | Through study completion; an average of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Eileen Hacker, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org